CLINICAL TRIAL: NCT04008251
Title: Treatment of Relapsed or Refractory B-cell Malignancies by Humanized CD19 Chimeric Antigen Receptor (CAR)-Modified T Cells
Brief Title: Humanized CD19 Chimeric Antigen Receptor (CAR)-Modified T Cell Therapy in Treating Patients With B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Sian Medical Technology Co., Ltd (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Jingzhou Central Hospital (Other); Xiangyang Central Hospital (Other); People Hospital Of Yichang (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-huCD19-01
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Acute Lymphoblastic Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second generation humanized CAR-T cells (Experimental): Patients receive humanized CD19 CAR-T cells transduced with a lentiviral vector on days 0/1/2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Genetic: Second generation humanized CAR-T cells

INTERVENTIONS:
Genetic: Second generation humanized CAR-T cells — Patients receive humanized CD19 CAR-T cells transduced with a lentiviral vector on days 0/1/2 in the absence of disease progression or unacceptable toxicity.

SUMMARY:
This is a single arm, open-label study to evaluate the safety and efficacy of humanized anti-CD19 CAR-T cells in patients with relapsed or refractory B cell Malignancies.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells (CAR-T cells) have the capabilities to recognize tumor associated antigen and kill tumor cells specifically. CAR-T therapy showed great effect on patients with relapsed or refractory B cell malignancies. To improve the efficacy and safety, the researchers designed a second-generation humanized CAR, consisting of humanized CD19 single chain variable fragment (scFv) and CD137 costimulatory domain. This study aims to evaluate the safety and effectiveness of humanized anti-CD19 CAR-T cells in patients with relapsed or refractory B cell Malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is pathologically and histologically confirmed as CD19 + B cell tumors, and has no effective treatment options currently, such as chemotherapy; or relapsed after auto-HSCT/allo-HSCT; or patients voluntarily choose CD19 CAR-T cells as a first treatment;
2. B cell hematological malignancies include the following three categories:

   A. B-cell acute lymphocytic leukemia (B-ALL);

   B. Indolent B-cell lymphoma (CLL, FL, MZL, LPL);

   C. Aggressive B-cell lymphoma (DLBCL, BL, MCL);
3. Aged from 14 to 70 years old;
4. Expected survival time > 6 months;
5. Female patients around childbearing age, negative pregnancy test before trial, and agreed to take effective contraceptive measures during the trial until the last visit;
6. Voluntarily participate in this experiment and sign informed consent by themself, or legally authorized representative.

Exclusion Criteria:

1. With a history of epilepsy or other central nervous system diseases;
2. Having graft-versus-host reaction, requires the use of immunosuppressants;
3. The presence of clinically significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within recent six months, or heart disease with cardiac function in any grade 3 (moderate) or 4 ( severe) (according to the New York Heart Association (NYHA) Functional Classification System);
4. Pregnant or lactating women (safety of this therapy for the unborn child is unknown);
5. Not curable active infection;
6. Patients with active hepatitis B or hepatitis C virus infection;
7. Combined use of systemic steroids within two weeks (except use of inhaled steroid recently or currently);
8. Using product of gene therapy before;
9. Creatinine> 2.5 mg / dl (221.0 umol/L); ALT / AST> 3 X the normal amount; Bilirubin> 2.0 mg / dl (34.2 umol/L);
10. Patients suffering from other uncontrolled diseases, and researchers believe that the patient is not suitable for trial;
11. Patients with HIV-infection;
12. Any situation that may increase the risk of patients or interfere with test results.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 5 years
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0)

SECONDARY OUTCOMES:
One-month remission rate | 1 month
  Response of B-ALL to CAR-T therapy was assessed on day 30 (±2), against the National Comprehensive Cancer Network (NCCN, Version 1.2015).
Overall survival | 5 years
  OS was calculated from the first CAR-T cell infusion to death or last follow-up (censored).
Event-free survival | 5 years
  EFS was calculated from the first CAR-T cell infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit (censored).
Relapse-free survival | 5 years
  RFS was calculated from the first CAR-T cell infusion to relapse or last visit (censored).
Rate of anti-CD19 CAR-T cells in bone marrow cells and peripheral blood cells | 5 years
  In vivo (bone marrow and peripheral blood) rate of CAR-T cells were determined by means of flow cytometry.
Quantity of anti-CD19 CAR-T cells in bone marrow cells and peripheral blood cells | 5 years
  In vivo (bone marrow and peripheral blood) quantity of CAR-T cells were determined by means of flow cytometry.
Quantity of anti-CD19 CAR copies in bone marrow cells and peripheral blood cells | 5 years
  In vivo (bone marrow and peripheral blood) quantity of anti-CD19 CAR copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Du M, Mayombo RTM, Liu J, Zhang Y, Liao D, Hu Y, Mei H. The impact of obesity and its related underlying diseases on cytokine release syndrome and the efficacy of CAR-T therapy in treating B-cell malignancies. Ann Hematol. 2025 Mar;104(3):1887-1895. doi: 10.1007/s00277-025-06338-6. Epub 2025 Apr 8. PMID 40195173
- [Derived] Zhang Y, Zhou F, Wu Z, Li Y, Li C, Du M, Luo W, Kou H, Lu C, Mei H. Timing of Tocilizumab Administration Under the Guidance of IL-6 in CAR-T Therapy for R/R Acute Lymphoblastic Leukemia. Front Immunol. 2022 Jun 21;13:914959. doi: 10.3389/fimmu.2022.914959. eCollection 2022. PMID 35799791